CLINICAL TRIAL: NCT06789172
Title: A Phase 1, Open-label, Multicenter, Dose-escalation and Cohort Expansion Study of OKN4395, a Triple Antagonist of EP2, EP4, and DP1 Prostanoid Receptors, as Monotherapy and in Combination With Pembrolizumab, in Patients With Advanced Solid Tumors
Brief Title: A Phase 1, First-in-human Study of OKN4395 and Pembrolizumab in Patients With Solid Tumors
Acronym: INVOKE
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Epkin (Industry)
Collaborators: Precision For Medicine (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OKN-4395-121
Record Dates: First submitted 2025-01-13; First posted 2025-01-23 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Solid Tumours; Sarcoma; HNSCC; Non Small Cell Lung Cancer; Head and Neck Squamous Cell Carcinoma; NSCLC; Pancreatic Adenocarcinoma; Colorectal Cancer (CRC); Myxofibrosarcoma (MFS); Solitary Fibrous Tumors; Dedifferentiated Liposarcoma; Undifferentiated Pleomorphic Sarcoma (UPS)
MeSH Terms: conditions — Sarcoma; Squamous Cell Carcinoma of Head and Neck; Carcinoma, Non-Small-Cell Lung; Colorectal Neoplasms; Dermatofibrosarcoma; Solitary Fibrous Tumors; Liposarcoma; Histiocytoma, Malignant Fibrous | interventions — pembrolizumab; Angptl4 protein, mouse; Histamine H2 Antagonists; Famotidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (9):
- Monotherapy Dose Escalation Phase (Phase 1a) (Experimental): The Monotherapy Escalation Phase will include increasing doses of OKN4395 alone in patients with solid tumors with a COX2-associated immunosuppressive pathway.
  Interventions: Drug: OKN4395
- Combination Dose Confirmation Phase (Phase 1a) (Experimental): The Combination Dose Confirmation Phase will include increasing or decreasing doses of OKN4395 in combination with pembrolizumab in patients with solid tumors with a COX2-associated immunosuppressive pathway. The first dose level used will be 1 level below the identified OBD/MTD for monotherapy. Subsequent dose levels tested will either be increased or decreased in response to observed toxicity.
  Interventions: Drug: OKN4395; Combination Product: Pembrolizumab
- Phase 1b Cohort 1: Sarcoma Food Effect (Fasted) (Experimental): Fasted first dose, and OBD/MTD (mono) dose of OKN4395 as monotherapy for the remainder of treatment.
  Interventions: Drug: OKN4395; Other: Fasting
- Phase 1b Cohort 1: Sarcoma Food Effect (Fed) (Experimental): Fed first dose, and OBD/MTD (mono) dose of OKN4395 as monotherapy for the remainder of treatment.
  Interventions: Drug: OKN4395; Other: Fed
- Phase 1b Cohort 2: Pancreas Gastric pH Effect (with H2RA) (Experimental): Co-administered H2RA (H2 receptor antagonist; famotidine) first dose, and OBD/MTD (mono) dose of OKN4395 as monotherapy for the remainder of treatment.
  Interventions: Drug: OKN4395; Drug: H2 Receptor Antagonist
- Phase 1b Cohort 2: Pancreas Gastric pH Effect (without H2RA) (Experimental): No co-administered H2RA (H2 receptor antagonist; famotidine) first dose, and OBD/MTD (mono) dose of OKN4395 as monotherapy for the remainder of treatment.
  Interventions: Drug: OKN4395
- Phase 1b Cohort 3: NSCLC (Experimental): OKN4395 (OBD/MTD combination dose) in combination with pembrolizumab
  Interventions: Drug: OKN4395; Combination Product: Pembrolizumab
- Phase 1b Cohort 4: Colorectal Cancer (Experimental): OKN4395 (OBD/MTD combination dose) in combination with pembrolizumab
  Interventions: Drug: OKN4395; Combination Product: Pembrolizumab
- Phase 1b Cohort 5: HNSCC (Experimental): OKN4395 (OBD/MTD combination dose) in combination with pembrolizumab
  Interventions: Drug: OKN4395; Combination Product: Pembrolizumab

INTERVENTIONS:
Drug: OKN4395 — OKN4395 oral dosing twice per day
Combination Product: Pembrolizumab — 200 mg IV every 3 weeks
  Arms: Combination Dose Confirmation Phase (Phase 1a); Phase 1b Cohort 3: NSCLC; Phase 1b Cohort 4: Colorectal Cancer; Phase 1b Cohort 5: HNSCC
Other: Fasting — Fasting before first dose of OKN4395
  Arms: Phase 1b Cohort 1: Sarcoma Food Effect (Fasted)
Other: Fed — Food provided to patient before first OKN4395 dose
  Arms: Phase 1b Cohort 1: Sarcoma Food Effect (Fed)
Drug: H2 Receptor Antagonist — Famotidine 20 mg IV (as a slow push over 2 minutes) administered 3 hours prior to OKN4395
  Other Names: Famotidine; H2RA
  Arms: Phase 1b Cohort 2: Pancreas Gastric pH Effect (with H2RA)

SUMMARY:
The purpose of this study is to investigate the study drug, OKN4395, administered alone and in combination with pembrolizumab.

The overall objectives of this study are to determine the safety and tolerability (degree to which side effects of a drug can be tolerated) of OKN4395 alone and in combination with pembrolizumab, OKN4395 and metabolites (broken-down substances) of OKN4395 levels in the blood, and antitumor activity of OKN4395 alone and in combination with pembrolizumab.

This study will be split into 2 parts. Part 1a will look at multiple doses of OKN4395 either alone (monotherapy) or with pembrolizumab (combination therapy) administered on day 1 of each 21-day cycle in patients with solid tumors until the participant has disease progression or discontinues for any reason. The dose of OKN4395 will be increased, after each group of 3 or more patients completes their first 3 weeks of treatment and their data is evaluated for safety, with a planned dose range from 10 mg twice a day to 450 mg twice a day through 13 dose levels. Part 1b will evaluate OKN4395 alone and in combination with pembrolizumab administered on day 1 of each 21-day cycle in patients with selected cancer types. Part 1b will comprise 5 cohorts: Cohort 1 in sarcoma (OKN4395 alone), Cohort 2 pancreatic adenocarcinoma (OKN4395 alone), Cohort 3 in non-small cell lung cancer (NSCLC), Cohort 4 in colorectal cancer, and Cohort 5 in head & neck squamous cell carcinoma (HNSCC), with cohorts 3 to 5 in combination with pembrolizumab. The monotherapy expansion Cohort 1 will also be used to explore the effect of food on the levels of OKN4395 in the blood. Similarly, Cohort 2 will be used to explore the effect of gastric pH on the levels of OKN4395 in the blood.

The overall study will enrol approximately 166 participants with up to 54 participants to receive OKN4395 alone and 12 participants to receive OKN4395 in combination with pembrolizumab in Part 1a, and 100 participants in Part 1b split: 40 on monotherapy and 60 on combination therapy. The study will be conducted in the US, Australia, UK and in the EU.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed disease, locally advanced or metastatic:

   For Phase 1a:

   Solid tumor with a COX2-associated immunosuppressive pathway, for which standard treatment options are not available, no longer effective, refused or not tolerated.

   For Phase 1b:

   For all cohorts, in the opinion of the investigator, all appropriate authorised treatment options should be exhausted
   * Cohort 1: Sarcoma (fibrous sarcoma [myxofibrosarcoma or solitary fibrous tumor], dedifferentiated liposarcoma, undifferentiated pleomorphic sarcoma or pleomorphic sarcoma), that is either refractory to or progressing on standard of care, with no more than 3 prior lines of systemic therapy. Patients with a solitary fibrous tumor can be included in the study without prior treatment if, in the investigator's opinion, it is in the participant's best interest and no established standard of care exists or is available.
   * Cohort 2: Pancreatic adenocarcinoma, with no more than 3 prior lines of systemic therapy. When known, KRAS and BRCA status should be provided.
   * Cohort 3: NSCLC (squamous or adenomatous without EGFR/ALK mutations), with previous platinum-based chemotherapy and a previous PD-(L)1 CPI regimen (unless not eligible/unwilling to receive such therapies), and no more than 3 prior lines of systemic therapy. When known, PD-L1 status should be provided.
   * Cohort 4: CRC (Microsatellite stable or Microsatellite instability - low), and no more than 4 prior lines of systemic therapy.
   * Cohort 5: HNSCC (oral cavity, oropharynx, larynx, hypopharynx), with a previous regimen containing a PD-(L)1 CPI (unless not eligible/unwilling to receive such therapies), and no more than 3 prior lines of systemic therapy. When known, PD-L1 and HPV status should be provided.
2. ECOG performance status of 0 or 1.
3. Recovery from any medically relevant AE/irAE from previous treatment regimen (defined as recovery to Grade ≤1 level per CTCAE v 5.0 before Screening, or chronic, stable, Grade 2 AEs [not worsened to Grade >2 for >3 months prior to screening]).
4. One or more new or growing tumor lesions amenable to a safe biopsy (at baseline, a suitable archival specimen obtained when not undergoing treatment and within 1 year [Phase 1a], or within 90 days and after the last administration of the previous systemic therapy [Phase 1b] is suitable). In addition (where applicable) an archival tumor biopsy collected before the start of the first-line treatment in the metastatic setting is requested (but optional).
5. At least one target lesion measurable by RECIST 1.1 as noted by local investigators/radiologists.
6. The ability to swallow and retain OKN4395 as an oral medication without significant gastrointestinal abnormalities that might alter absorption.
7. The willingness and ability to comply with the food effect (Phase 1b Cohort 1), or gastric pH effect (Phase 1b Cohort 2) evaluation randomizations and requirements.
8. Adequate hematologic, renal, and hepatic function (based on local laboratory assessments):

   1. Hematological variables: absolute neutrophil counts ≥1.5 × 109 /L, platelet counts ≥75 × 109 /L, and hemoglobin ≥8 g/dL
   2. Renal variables: creatinine clearance ≥ 60 mL/min1
   3. Hepatic variables: total serum bilirubin ≤1.5 × ULN, AST and ALT ≤3 × ULN, and ALP ≤2.5 × ULN; except for hyperbilirubinemia of Gilbert's syndrome (participants with Gilbert's syndrome can be included if total serum bilirubin ≤5× ULN and direct bilirubin ≤1.5 x ULN)
   4. Serum albumin ≥30 g/L

Exclusion Criteria:

1. Ongoing or recent anticancer therapy within the following timeframe prior to first dose of study drug:

   1. Chemotherapy, ADCs, or other antibodies < 21 days
   2. Immunotherapy or cellular therapy < 28 days
   3. Radiation therapy (palliative radiation for bone pain <48 hours; stereotactic or small field brain irradiation <7 days; all other radiation therapy <14 days)
   4. TKI or any other anticancer therapy < 5 half-lives or < 7 days, whichever is longer
2. Central nervous system metastasis (radiologically progressive, or clinically symptomatic, or requiring immunosuppressive therapies [including low dose steroids]).
3. Any active infection (bacterial, viral, fungal) requiring IV systemic therapy.
4. Unstable COPD defined as frequent or severe exacerbations per investigator discretion.
5. Known active HBV or HCV infection or positive test(s) as per CDC guidance (Centers for Disease Control and Prevention, 2023, 2024) or HIV infection with CD4 lymphocyte count <350 cells/μL at time of Screening, or failure to achieve and maintain virologic suppression defined as confirmed HIV RNA level < 50 or lower limit of detection by the local available assay at time of Screening and for at least 12 weeks prior to Screening. No testing is required unless medically indicated or mandated by local authorities.
6. Known history of bleeding disorders, INR ≥1.5 × ULN at screening (or INR and/or aPTT within therapeutic range if on anticoagulation therapy), or a history of gastrointestinal bleeding (inflammatory, ulcerative, or diverticular) within the last 2 years.
7. Known H. pylori infection without proof of eradication at least 2 months prior to screening.
8. Systemic treatment with any drug known to impact gastrointestinal pH within 7 days (PPIs) or 12 hours (H2 antagonists) of first dose of OKN4395.
9. Acute treatment with any systemic steroid therapy (>10 mg prednisone equivalent), or any corticosteroid medication within 14 days of first dose of OKN4395 for any condition.
10. For participants planned to receive combination therapy: Ongoing and history of active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Any replacement therapy (i.e. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment and is allowed. Participants with hyperthyroidism or hypothyroidism but that are stable on hormone replacement are also allowed.
11. Systemic treatment with NSAIDs, COX2 inhibitors, or synthetic prostaglandins within 5 half-lives prior to the first dose of OKN4395 (acetylsalicylic acid ≤ 160 mg/day, or 325 mg ≤ 3 times/week is permitted).
12. Systemic treatment with strong inhibitors/inducers of CYP and UGT enzymes within 14 days of first dose of OKN4395.
13. QTcF interval of > 450 ms based on mean of the central triplicate readings.
14. Known hypersensitivity to any excipients of the OKN4395 formulation or pembrolizumab (for combination cohorts).
15. Pregnant or lactating women. Women of childbearing potential must have a negative serum pregnancy test at screening and have a negative a urine dipstick pregnancy test prior to the initiation of study treatment (can be done on C1-D1 visit).
16. Evidence of any other active malignancy requiring systemic therapy within the 2 years prior to Screening. (Exceptions: non-melanoma skin cancer, in situ melanoma, in situ cervical cancer, ductal carcinoma in situ of the breast, or localized and presumed cured prostate cancer; participants on long-term anti-hormonal therapy for a prior malignancy are allowed if the malignancy has not been active within the prior 2 years).
17. History or current evidence of any condition, surgical or medical therapy, or laboratory abnormalities that might confound the results of the study, make study drug administration hazardous, interfere with the participant's involvement for the full duration of the study, or make it difficult to monitor AEs such that, in the opinion of the treating physician, it is not in the best interest of the participant to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Estimated)
Dates: Start 2025-01-23 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of DLTs in participants treated with OKN4395 as monotherapy and in combination with pembrolizumab. (Phase 1a) | From enrolment of the first participant until the end of Phase 1a or until the DLT threshold is reached; up to 27 months
  DLTs = dose-limiting toxicities
Incidence and severity of TEAEs in participants treated with OKN4395 as a monotherapy and in combination with pembrolizumab in solid tumors. (Phase 1a) | From enrolment of the first participant to the end of Phase 1a; up to 27 months
  TEAEs = treatment-emergent adverse events
Incidence and severity of SAEs in participants treated with OKN4395 as a monotherapy and in combination with pembrolizumab in solid tumors. (Phase 1a) | From enrolment of the first participant to the end of Phase 1a; up to 27 months
  SAEs = serious adverse events
Incidence of dose interruptions, dose reductions, and dose intensities in participants treated with OKN4395 as a monotherapy and in combination with pembrolizumab in solid tumors. (Phase 1a) | From enrolment of the first participant to the end of Phase 1a; up to 27 months
Incidence and severity of clinically relevant ECG abnormalities in participants treated with OKN4395 as a monotherapy and in combination with pembrolizumab in solid tumors. (Phase 1a) | From enrolment of the first participant to the end of Phase 1a; up to 27 months
  ECG = electrocardiogram
Incidence and severity of laboratory abnormalities in participants treated with OKN4395 as a monotherapy and in combination with pembrolizumab in solid tumors. (Phase 1a) | From enrolment of the first participant to the end of Phase 1a; up to 27 months
  Graded where appropriate with the CTCAE v5.0.
Incidence and severity of clinically relevant changes in vital signs in participants treated with OKN4395 as a monotherapy and in combination with pembrolizumab in solid tumors. (Phase 1a) | From enrolment of the first participant to the end of Phase 1a; up to 27 months
To assess the overall response rate in participants treated with OKN4395 as monotherapy and in combination with pembrolizumab in selected cancer types. (Phase 1b) | From enrolment of first participant in Phase 1b until 24 weeks after the last participant is enrolled in Phase 1b; up to 12 months from beginning of Phase 1b

SECONDARY OUTCOMES:
To assess the overall response rate in participants treated with OKN4395 as monotherapy and in combination with pembrolizumab in selected cancer types. (Phase 1a) | From enrolment of the first participant until the end of Phase 1a or until the DLT threshold is reached; up to 27 months
To assess the disease control rate at >=12 weeks in participants treated with OKN4395 as monotherapy and in combination with pembrolizumab in selected cancer types. (Phase 1a) | From enrolment of the first participant until the end of Phase 1a or until the DLT threshold is reached; up to 27 months
To assess the duration of response in participants treated with OKN4395 as monotherapy and in combination with pembrolizumab in selected cancer types. (Phase 1a) | From enrolment of the first participant until the end of Phase 1a or until the DLT threshold is reached; up to 27 months
To assess the progression-free survival in participants treated with OKN4395 as monotherapy and in combination with pembrolizumab in selected cancer types. (Phase 1a) | From enrolment of the first participant until the end of Phase 1a or until the DLT threshold is reached; up to 27 months
To assess the time to treatment failure in participants treated with OKN4395 as monotherapy and in combination with pembrolizumab in selected cancer types. (Phase 1a) | From enrolment of the first participant until the end of Phase 1a or until the DLT threshold is reached; up to 27 months
To assess the overall survival rate at 24 weeks in participants treated with OKN4395 as monotherapy and in combination with pembrolizumab in selected cancer types. (Phase 1a) | From enrolment of the first participant until the end of Phase 1a or until the DLT threshold is reached; up to 27 months
To characterize the maximum plasma concentration (pharmacokinetics) of OKN4395 and its AG metabolite. (Phase 1a) | From enrolment of the first participant until the end of Phase 1a or until the DLT threshold is reached; up to 27 months
To characterize the area under the curve (pharmacokinetics) of OKN4395 and its AG metabolite. (Phase 1a) | From enrolment of the first participant until the end of Phase 1a or until the DLT threshold is reached; up to 27 months
To characterize the terminal half life (pharmacokinetics) of OKN4395 and its AG metabolite. (Phase 1a) | From enrolment of the first participant until the end of Phase 1a or until the DLT threshold is reached; up to 27 months
To characterize the clearance (pharmacokinetics) of OKN4395 and its AG metabolite. (Phase 1a) | From enrolment of the first participant until the end of Phase 1a or until the DLT threshold is reached; up to 27 months
To characterize the accumulation index (pharmacokinetics) of OKN4395 and its AG metabolite. (Phase 1a) | From enrolment of the first participant until the end of Phase 1a or until the DLT threshold is reached; up to 27 months
To assess the disease control rate at >=12 weeks in participants treated with OKN4395 as monotherapy and in combination with pembrolizumab in selected cancer types. (Phase 1b) | From enrolment of first participant in Phase 1b until 24 weeks after the last participant is enrolled in Phase 1b; up to 12 months from beginning of Phase 1b
To assess the duration of response in participants treated with OKN4395 as monotherapy and in combination with pembrolizumab in selected cancer types. (Phase 1b) | From enrolment of first participant in Phase 1b until 24 weeks after the last participant is enrolled in Phase 1b; up to 12 months from beginning of Phase 1b
To assess the progression-free survival in participants treated with OKN4395 as monotherapy and in combination with pembrolizumab in selected cancer types. (Phase 1b) | From enrolment of first participant in Phase 1b until 24 weeks after the last participant is enrolled in Phase 1b; up to 12 months from beginning of Phase 1b
To assess the time to treatment failure in participants treated with OKN4395 as monotherapy and in combination with pembrolizumab in selected cancer types. (Phase 1b) | From enrolment of first participant in Phase 1b until 24 weeks after the last participant is enrolled in Phase 1b; up to 12 months from beginning of Phase 1b
To assess the overall survival rate at 24 weeks in participants treated with OKN4395 as monotherapy and in combination with pembrolizumab in selected cancer types. (Phase 1b) | From enrolment of first participant in Phase 1b until 24 weeks after the last participant is enrolled in Phase 1b; up to 12 months from beginning of Phase 1b
Incidence and severity of TEAEs in participants treated with OKN4395 as a monotherapy and in combination with pembrolizumab in solid tumors. (Phase 1b) | From enrolment of first participant in Phase 1b until 24 weeks after the last participant is enrolled in Phase 1b; up to 12 months from beginning of Phase 1b
Incidence and severity of SAEs in participants treated with OKN4395 as a monotherapy and in combination with pembrolizumab in solid tumors. (Phase 1b) | From enrolment of first participant in Phase 1b until 24 weeks after the last participant is enrolled in Phase 1b; up to 12 months from beginning of Phase 1b
Incidence of dose interruptions, dose reductions, and dose intensities in participants treated with OKN4395 as a monotherapy and in combination with pembrolizumab in solid tumors. (Phase 1b) | From enrolment of first participant in Phase 1b until 24 weeks after the last participant is enrolled in Phase 1b; up to 12 months from beginning of Phase 1b
To characterize the maximum plasma concentration (pharmacokinetics) of OKN4395 and its AG metabolite. (Phase 1b) | From enrolment of first participant in Phase 1b until 24 weeks after the last participant is enrolled in Phase 1b; up to 12 months from beginning of Phase 1b
Incidence and severity of clinically relevant ECG abnormalities in participants treated with OKN4395 as a monotherapy and in combination with pembrolizumab in solid tumors. (Phase 1b) | From enrolment of first participant in Phase 1b until 24 weeks after the last participant is enrolled in Phase 1b; up to 12 months from beginning of Phase 1b
Incidence and severity of laboratory abnormalities in participants treated with OKN4395 as a monotherapy and in combination with pembrolizumab in solid tumors. (Phase 1b) | From enrolment of first participant in Phase 1b until 24 weeks after the last participant is enrolled in Phase 1b; up to 12 months from beginning of Phase 1b
Incidence and severity of clinically relevant changes in vital signs in participants treated with OKN4395 as a monotherapy and in combination with pembrolizumab in solid tumors. (Phase 1b) | From enrolment of first participant in Phase 1b until 24 weeks after the last participant is enrolled in Phase 1b; up to 12 months from beginning of Phase 1b
To characterize the area under the curve (pharmacokinetics) of OKN4395 and its AG metabolite. (Phase 1b) | From enrolment of first participant in Phase 1b until 24 weeks after the last participant is enrolled in Phase 1b; up to 12 months from beginning of Phase 1b
To characterize the terminal half life (pharmacokinetics) of OKN4395 and its AG metabolite. (Phase 1b) | From enrolment of first participant in Phase 1b until 24 weeks after the last participant is enrolled in Phase 1b; up to 12 months from beginning of Phase 1b
To characterize the clearance (pharmacokinetics) of OKN4395 and its AG metabolite. (Phase 1b) | From enrolment of first participant in Phase 1b until 24 weeks after the last participant is enrolled in Phase 1b; up to 12 months from beginning of Phase 1b
To characterize the accumulation index (pharmacokinetics) of OKN4395 and its AG metabolite. (Phase 1b) | From enrolment of first participant in Phase 1b until 24 weeks after the last participant is enrolled in Phase 1b; up to 12 months from beginning of Phase 1b

CONTACTS AND LOCATIONS:
Locations (10):
- United States (3):
  - Precision NextGen Oncology and Research Center, Beverly Hills, California
  - Sarcoma Oncology Center, Santa Monica, California
  - MD Anderson Cancer Center, Houston, Texas
- Australia (2):
  - Chris O'Brien Lifehouse, Sydney, New South Wales
  - Linear Clinical Research, Perth, Western Australia
- United Kingdom (5):
  - The Beatson, Glasgow
  - Leicester Royal Infirmary, Leicester
  - University College London Hospital, London
  - The Christie, Manchester
  - Churchill Hospital, Oxford

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Information about the INVOKE trial — https://www.epkin.ai/invoke-trial
- See also: Information for participants in the INVOKE trial — https://www.epkin.ai/participant-information